CLINICAL TRIAL: NCT02236650
Title: A Pilot Study of Primary Care Stepping Stones Triple P for Children With Autism
Brief Title: Primary Care Stepping Stones Triple P for Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Debra H. Zand, Ph.D., Associate Professor of Pediatrics, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLUBM_24272
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Autism
Keywords: Parental Resilience; Parental Stress; Family Adaptation; Autistic Disorder; Behavior; Child Behavior; Child Development Disorders; Pervasive Developmental Disabilities; Caregivers; Parents; Parenting; Primary Health Care
MeSH Terms: conditions — Autistic Disorder; Behavior; Child Behavior; Developmental Disabilities | interventions — (tris(diphenylphosphinomethyl)phenylborate)(p-tolylnitrido)iron(I); Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary Care Stepping Stones Triple P (Experimental): Primary Care Stepping Stones Triple P program (PC-SS Triple P) - a parenting and family support strategy that aims to prevent and treat behavioral problems in children by enhancing parental resilience.
  Interventions: Behavioral: Primary Care Stepping Stones Triple P (PC-SS Triple P)
- Wait List Control (WLC) (Active Comparator): Wait List Control - Participants who will have access to treatment as usual services during the 4 weeks between baseline and 4 week assessment time points and then will have the opportunity to receive PC-SS Triple P.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Primary Care Stepping Stones Triple P (PC-SS Triple P) — PC-SS Triple P is a parenting and family support strategy that aims to prevent and treat behavioral problems in children by enhancing parental resilience.
  Other Names: Postive Parenting Program; Triple P; Stepping Stones Triple P; Stepping Stones Positive Parenting Program
  Arms: Primary Care Stepping Stones Triple P
Other: Treatment as Usual — Treatment as Usual for 4 weeks
  Other Names: Service as Usual
  Arms: Wait List Control (WLC)

SUMMARY:
The purpose of this study is to determine the effectiveness of Primary Care Stepping Stones Triple P (PC-SS Triple P), an empirically supported parent mediated intervention, to improve the behavioral functioning of children newly diagnosed with Autism (aged 2-12 years), increase parental resilience and decrease parental stress.

DETAILED DESCRIPTION:
Research literature exists on best practices for screening and diagnosing children with Autism. However, less is known about how to intervene with the child's parent. Across studies, relative to parents of children without disabilities, parents of children with Autism have reported higher levels of stress and lower levels of parenting competence. Such stress places children at risk for adverse developmental outcomes

The proposed study aims to determine the effectiveness of Primary Care Stepping Stones Triple P (PC-SS Triple P), an empirically supported parent mediated intervention, to improve the behavioral functioning of children newly diagnosed with Autism (aged 2-12 years), increase parental resilience and decrease parental stress.

The specific hypotheses include:

1. Children whose parents receive PC-SS Triple P will demonstrate significantly greater improvements in their behavioral functioning than children of parents receiving Wait-list Control (WLC) at service closure.
2. At service closure, parents receiving the PC-SS Triple P intervention will be more resilient and demonstrate lower levels of stress than parents in the Wait-List Control (WLC) condition.
3. Parenting resilience and levels of parental stress will be positively associated with improvements in child behavior.

Seventy-six parents of children newly diagnosed with Autism will be randomized into one of two conditions: a) PC-SS Triple P (N=38) or b) Wait List Control (WLC; N=38). Study data will be collected with the assistance of a data collector appropriately trained in human subject rights protections.

It is anticipated that the present project will assist in the development and use of evidence-based practices for working with parents of children newly diagnosed with Autism within pediatric settings.

ELIGIBILITY:
Inclusion Criteria:

Parent inclusion criteria:

* being at least 18 years of age

Index child inclusion criteria:

* receives a Diagnostic and Statistical Manual V (DSM-V) diagnosis of Autism with mild or moderate severity within 12 months of study onset.
* age is > or equal to 24 months (2 years, 0 months) and < or equal to 155 months old (12 years, 11 months).

Exclusion Criteria:

Parent exclusion criteria:

* inability to provide informed consent.
* being non-English speaking.

Index child exclusion criteria:

* being a ward of the State of Missouri.
* being a sibling of another study participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Eyberg Child Behavior Inventory Score at 4 weeks | Baseline and 4 weeks
  Measure conduct problem behavior in children between the ages of 2 and 16 years.
Change from Baseline in Connor-Davidson Resilience Scale Score at 4 weeks | Baseline and 4 weeks
  General scale of resilience in adult populations with a bias towards coping with stress and adversity.
Change from Baseline in Parent Stress Index - Short Form Score at 4 weeks | Baseline and 4 weeks
  Sources and different types of stress that every parent can experience. Provides information in 4 specific domains of parenting stress:
  1. Parental Distress,
  2. Parent-Child Dysfunctional Interaction,
  3. Difficult Child, and
  4. Total Stress.
Change from Baseline in Family Assessment Device score at 4 weeks | Baseline and 4 weeks
  Assesses family functioning on six different dimensions:
  1. Problem Solving (ability to resolve problems),
  2. Communication (exchange of clear and direct verbal information),
  3. Roles (division of responsibility for completing family tasks),
  4. Affective Responsiveness (ability to respond with appropriate emotion),
  5. Affective Involvement (degree to which family members are involved and interested in one another), and
  6. Behavior Control (manner used to express and maintain standards of behavior).

SECONDARY OUTCOMES:
Change from Baseline in Aberrant Behavior Checklist Score at 4 weeks | Baseline and 4 weeks
  Assesses behavior problems in individuals with developmental disabilities across 5 domains:
  1. Irritability and Agitation (15 items)
  2. Lethargy and Social Withdrawal (16 items)
  3. Stereotypic Behavior (7 items)
  4. Hyperactivity and Noncompliance (16 items) and
  5. Inappropriate Speech (4 items).
Change from Baseline in The Parenting Scale Score at 4 weeks | Baseline and 4 weeks
  Measures dysfunctional discipline styles in parents by asking about the probability with which the parent uses particular discipline strategies. It yields four scores:
  1. Total score,
  2. Laxness (permissive, inconsistent discipline);
  3. Over-reactivity (harsh, emotional, authoritarian discipline and irritability); and
  4. Verbosity/Hostility (use of verbal or physical force).
Change from Baseline in the Parenting Sense of Competence Scale Score at 4 weeks | Baseline and 4 weeks
  Measures parents' sense of confidence and satisfaction with their parenting and their self-efficacy in the parenting role.

CONTACTS AND LOCATIONS:
Overall Officials: Debra H. Zand, PhD, Principal Investigator — Saint Louis University School of Medicine, Department of Pediatrics, Division of Developmental Pediatrics
Locations (1):
- Saint Louis University, Knights of Columbus Developmental Center, St Louis, Missouri, United States

REFERENCES:
- [Background] Turner K, Markie-Dadds C, Sanders M. Practitioner's manual for primary care tripleP. Brisbane, QLD, Australia: Triple P International Pty. Ltd.; 2010.
- [Background] Mazzucchelli T, Sanders M. Stepping Stones Triple P: A Population Approach to the Promotion of Competent Parenting of Children with Disability. Brisbane, Queensland, Australia,: The University of Queensland;2012.
- [Background] Prinz RJ, Sanders MR, Shapiro CJ, Whitaker DJ, Lutzker JR. Population-based prevention of child maltreatment: the U.S. Triple p system population trial. Prev Sci. 2009 Mar;10(1):1-12. doi: 10.1007/s11121-009-0123-3. PMID 19160053
- [Background] Sanders M, Morawska A. Can changing parental knowledge, dysfunctional expectations and attributions, and emotion regulation improve outcomes for children? In: Tremblay R, Boivin M, Peters R, eds. Encyclopedia on Early Childhood Development [online]. 2nd ed. Montreal, Quebec: Centre of Excellence for Early Childhood Development 2008:1-12.
- [Background] Sanders MR, Markie-Dadds C, Tully LA, Bor W. The triple P-positive parenting program: a comparison of enhanced, standard, and self-directed behavioral family intervention for parents of children with early onset conduct problems. J Consult Clin Psychol. 2000 Aug;68(4):624-40. PMID 10965638
- [Background] Sanders, Mazzucchelli T, Studman L. Stepping Stones Triple P: The theoretical basis and development of an evidence-based positive parenting program for families with a child who has a disability. Journal of Intellectual & Developmental Disability. 2004 2004;29(3):265-283.
- [Background] Tellegen CL, Sanders MR. Stepping Stones Triple P-Positive Parenting Program for children with disability: a systematic review and meta-analysis. Res Dev Disabil. 2013 May;34(5):1556-71. doi: 10.1016/j.ridd.2013.01.022. Epub 2013 Mar 6. PMID 23475006
- [Background] Whittingham K, Sofronoff K, Sheffield J, Sanders MR. Stepping Stones Triple P: an RCT of a parenting program with parents of a child diagnosed with an autism spectrum disorder. J Abnorm Child Psychol. 2009 May;37(4):469-80. doi: 10.1007/s10802-008-9285-x. PMID 19023654
- [Background] Becvar D. Handbook of family resilience. New York, NY: Springer; 2012.
- [Background] Roberts C, Mazzucchelli T, Studman L, Sanders MR. Behavioral family intervention for children with developmental disabilities and behavioral problems. J Clin Child Adolesc Psychol. 2006 Jun;35(2):180-93. doi: 10.1207/s15374424jccp3502_2. PMID 16597214
- [Background] Eyberg S, Pincus D. Eyberg Child Behavior Inventory and Sutter-Eyberg Student Behaviour Inventory- Revised: Professional manual. Odessa, FL: Psychological Assessment Resources; 1999.
- [Background] Aman MG, Singh NN, Stewart AW, Field CJ. The aberrant behavior checklist: a behavior rating scale for the assessment of treatment effects. Am J Ment Defic. 1985 Mar;89(5):485-91. PMID 3993694
- [Background] Karabekiroglu K, Aman MG. Validity of the aberrant behavior checklist in a clinical sample of toddlers. Child Psychiatry Hum Dev. 2009 Mar;40(1):99-110. doi: 10.1007/s10578-008-0108-7. Epub 2008 Jul 4. PMID 18600444
- [Background] Guy WR, 1976. M. ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: US Department of Heath, Education, and Welfare, Public Health Service, Alcohol, Drug Abuse, and Mental Health Administration; 1976.
- [Background] Arnold D, O'Leary S, Wolff S, Acher M. The Parenting Scale: A measure of dysfunctional parenting in discipline situations. Psychological Assessment. 1993 1993;5:137-144.
- [Background] Johnston C, Mash E. A measure of parenting satisfaction and efficacy. Journal of Clinical Child Psychology. 1989 1989;18:167-175.
- [Background] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Andrews G, Slade T. Interpreting scores on the Kessler Psychological Distress Scale (K10). Aust N Z J Public Health. 2001 Dec;25(6):494-7. doi: 10.1111/j.1467-842x.2001.tb00310.x. PMID 11824981
- [Background] Kessler RC, Barker PR, Colpe LJ, Epstein JF, Gfroerer JC, Hiripi E, Howes MJ, Normand SL, Manderscheid RW, Walters EE, Zaslavsky AM. Screening for serious mental illness in the general population. Arch Gen Psychiatry. 2003 Feb;60(2):184-9. doi: 10.1001/archpsyc.60.2.184. PMID 12578436
- [Background] Abidin R. Parent Stress Index-Short Form. Florida: Psychological Assessment Resources Incorporated; 1995.
- [Background] Zaidman-Zait A, Mirenda P, Zumbo BD, Wellington S, Dua V, Kalynchuk K. An item response theory analysis of the Parenting Stress Index-Short Form with parents of children with autism spectrum disorders. J Child Psychol Psychiatry. 2010 Nov;51(11):1269-77. doi: 10.1111/j.1469-7610.2010.02266.x. PMID 20546082
- [Background] Thomas KC, Ellis AR, McLaurin C, Daniels J, Morrissey JP. Access to care for autism-related services. J Autism Dev Disord. 2007 Nov;37(10):1902-12. doi: 10.1007/s10803-006-0323-7. Epub 2007 Mar 19. PMID 17372817
- [Background] Aitken L, Gallagher R, Madronio C. Principles of recruitment and retention in clinical trials. Int J Nurs Pract. 2003 Dec;9(6):338-46. doi: 10.1046/j.1440-172x.2003.00449.x. PMID 14984070
- [Background] Lovato LC, Hill K, Hertert S, Hunninghake DB, Probstfield JL. Recruitment for controlled clinical trials: literature summary and annotated bibliography. Control Clin Trials. 1997 Aug;18(4):328-52. doi: 10.1016/s0197-2456(96)00236-x. PMID 9257072
- [Background] Meneses K, Roche C. Recruitment and retention in clinical research. Perioperative Nursing Clinics. 2009;4:259-268.
- [Background] Bethell CD, Read D, Neff J, Blumberg SJ, Stein RE, Sharp V, Newacheck PW. Comparison of the children with special health care needs screener to the questionnaire for identifying children with chronic conditions--revised. Ambul Pediatr. 2002 Jan-Feb;2(1):49-57. doi: 10.1367/1539-4409(2002)0022.0.co;2. PMID 11888438
- [Background] Sandelowski M. Whatever happened to qualitative description? Res Nurs Health. 2000 Aug;23(4):334-40. doi: 10.1002/1098-240x(200008)23:43.0.co;2-g. PMID 10940958
- [Background] Sandelowski M. What's in a name? Qualitative description revisited. Res Nurs Health. 2010 Feb;33(1):77-84. doi: 10.1002/nur.20362. PMID 20014004
- [Background] Faul F, Erdfelder E, Buchner A, Lang AG. Statistical power analyses using G*Power 3.1: tests for correlation and regression analyses. Behav Res Methods. 2009 Nov;41(4):1149-60. doi: 10.3758/BRM.41.4.1149. PMID 19897823
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Baron RM, Kenny DA. The moderator-mediator variable distinction in social psychological research: conceptual, strategic, and statistical considerations. J Pers Soc Psychol. 1986 Dec;51(6):1173-82. doi: 10.1037//0022-3514.51.6.1173. PMID 3806354
- [Background] Judd C, Kenny D. Process analysis: Estimating mediation in treatment evaluations. Evaluation Review. 1981;5:602-619.
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of Autism Spectrum Disorders Autism and Developmental Disabilities Monitoring Network, 14 Sites in the United States. Atlanta, GA: Centers for Disease Control,; 2002.
- [Background] Yeargin-Allsopp M, Rice C, Karapurkar T, Doernberg N, Boyle C, Murphy C. Prevalence of autism in a US metropolitan area. JAMA. 2003 Jan 1;289(1):49-55. doi: 10.1001/jama.289.1.49. PMID 12503976
- [Background] Drew A, Baird G, Baron-Cohen S, Cox A, Slonims V, Wheelwright S, Swettenham J, Berry B, Charman T. A pilot randomised control trial of a parent training intervention for pre-school children with autism. Preliminary findings and methodological challenges. Eur Child Adolesc Psychiatry. 2002 Dec;11(6):266-72. doi: 10.1007/s00787-002-0299-6. PMID 12541005
- [Background] Blandon AY, Calkins SD, Keane SP. Predicting emotional and social competence during early childhood from toddler risk and maternal behavior. Dev Psychopathol. 2010 Winter;22(1):119-32. doi: 10.1017/S0954579409990307. PMID 20102651
- [Background] McConachie H, Diggle T. Parent implemented early intervention for young children with autism spectrum disorder: a systematic review. J Eval Clin Pract. 2007 Feb;13(1):120-9. doi: 10.1111/j.1365-2753.2006.00674.x. PMID 17286734
- [Background] Oosterling I, Visser J, Swinkels S, Rommelse N, Donders R, Woudenberg T, Roos S, van der Gaag RJ, Buitelaar J. Randomized controlled trial of the focus parent training for toddlers with autism: 1-year outcome. J Autism Dev Disord. 2010 Dec;40(12):1447-58. doi: 10.1007/s10803-010-1004-0. PMID 20440639
- [Background] Developmental surveillance and screening of infants and young children. Pediatrics. 2001 Jul;108(1):192-6. doi: 10.1542/peds.108.1.192. PMID 11433077
- See also: Family Research Collaborative - Autism & Parenting Resilience — https://sites.google.com/a/slu.edu/debra-h-zand-ph-d/parent-child-intervention-research-team-p-chirt